CLINICAL TRIAL: NCT04815408
Title: A Phase II Study of PD-1 Antibody Plus Neoadjuvant Chemotherapy for Advanced-stage Ovarian Cancer (Z2HOC-01)
Brief Title: PD-1 Antibody Combined Neoadjuvant Chemotherapy for Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Z2HOC-01
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer; Neoadjuvant Chemotherapy; Anti-PD-1; Neoadjuvant Immunotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — tislelizumab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIC (Experimental): 1. Neoadjuvant treatment BGB-A317 200mg q3 weeks (total 3 dosing) Chemotherapy regimen: albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5 q3 weeks (total 3 dosing)
  2. Interval debulking surgery and HIPEC
  3. Adjuvant treatment Chemotherapy regimen: albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5, Bevacizumab 7.5mg/kg q3 weeks (total 3 dosing)
  Interventions: Drug: BGB-A317; Drug: albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5
- NC (Active Comparator): 1. Neoadjuvant treatment Chemotherapy regimen: albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5 q3 weeks (total 3 dosing)
  2. Interval debulking surgery and HIPEC
  3. Adjuvant treatment Chemotherapy regimen: albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5, Bevacizumab 7.5mg/kg q3 weeks (total 3 dosing)
  Interventions: Drug: albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5

INTERVENTIONS:
Drug: BGB-A317 — PD-1 antibody，Tislelizumab (BGB-A317)
  Arms: NIC
Drug: albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5 — albumin-bound paclitaxel 260mg/m2 , Carboplatin AUC 5

SUMMARY:
The main purpose of this study is to validate the efficacy and safety of anti-PD-1 in combination with neoadjuvant chemotherapy in women with advanced ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of ovary, fallopian tube, primary peritoneum (Non-mucinous adenocarcinoma)
2. Clinical stage IIIC/IV, and IIIC with Suidan CT ≥3 or Fagotti ≥8
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 ~ 2
4. Not received any immunotherapy before
5. Willing to participate in this study, and sign the informed consent.

Exclusion Criteria:

1. With other uncontrolled malignant tumors.
2. Any disease requiring systemic treatment with a corticosteroid (prednisone or equivalent daily dose of > 10mg) or other immunosuppressive agents during the 14 days prior to randomization.The use of topical substitute steroids (daily dose ≤10mg of prednisone or its equivalent) and prescription corticosteroids for short-term (≤7 days) prophylactic use or for the treatment of non-autoimmune conditions is permitted.Has any active autoimmune disease or a history of autoimmunity.
3. A history of active autoimmune disease or autoimmune disease that may recur.Enrolment was allowed for well-controlled type 1 diabetes, hypothyroidism requiring only hormone replacement therapy, well-controlled celiac disease, skin conditions (such as vitiligo, psoriasis, or alopecia) that did not require systemic treatment, or conditions that were not expected to recede without an external cause.
4. A history of interstitial lung disease, non-infectious pneumonia, or poorly controlled diseases (including pulmonary fibrosis, acute lung disease, etc.).
5. Subjects with active hepatitis B (defined as positive hepatitis B virus surface antigen [HBsAg] test result and HBV-DNA test value higher than the upper limit of normal value in the laboratory of the research center) or hepatitis C (defined as positive hepatitis C virus surface antibody [HCSAB] test result and positive HCV-RNA test result).
6. Known human immunodeficiency virus (HIV) infection (known to be HIV positive).
7. Have received live vaccine within 30 days before the first administration.This includes but is not limited to the following: mumps, rubella, measles, varicella/herpes zoster (varicella), yellow fever, rabies, BCG and typhoid vaccines (inactivated virus vaccines are allowed).
8. With uncontrolled cardiac clinical symptoms or diseases.
9. Allergic to any drug in this program.
10. At the discretion of the Investigator, the subject has a history or current evidence of any disease, treatment or laboratory anomaly that may confuse the results, interfere with the participants' participation throughout the study, or is not in the best interest of the participants to participate in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 12 months
  12 months progression-free survival rate will be estimated, and 95% confidence intervals will be calculated.

SECONDARY OUTCOMES:
R0 rate | after interval debulking surgery for one week
  R0 rate of IDS(interval debulking surgery) after neoadjuvant chemotherapy(after the completion of 3rd cycle)
CRR | 3 months
  CRR is defined as the percentage of the participants in the ITT population who have a Complete Response or Partial Response. The CRR will be assessed by a blind independent central reviewer per RECIST 1.1
PRR | 3 months
  At interval cytoreduction pathologic complete remission rate will be measured using RECIST and immune-related response criteria.
OS | 5 years
  OS is defined as the time from the date of randomization until death.
AEs | 3 months
  Proportion of patients with grade 3 or more treatment-related adverse events(except hematologic toxicity) graded by CTCAE v5 in neoadjuvant chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Jianwei Zhou, MD, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhu Y, Fei J, Zhu X, Zhang J, Zhou J, Zhang Z. Efficacy and safety of NeoAdjuvant chemotherapy with or without tIslelizumab followed by debulking surgery for oVarian cancEr (NAIVE study) in China: study protocol of an open-label, phase II, randomised controlled trial. BMJ Open. 2025 Feb 5;15(2):e092545. doi: 10.1136/bmjopen-2024-092545. PMID 39909529